CLINICAL TRIAL: NCT03873805
Title: A Phase I Study to Evaluate PSCA-Targeting Chimeric Antigen Receptor (CAR)-T Cells for Patients With PSCA+ Metastatic Castration Resistant Prostate Cancer
Brief Title: PSCA-CAR T Cells in Treating Patients With PSCA+ Metastatic Castration Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17483; NCI-2019-01264 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17483 (Other: City of Hope Medical Center)
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (PSCA CAR T cells) (Experimental): Patients may receive lymphodepleting regimen (either standard or modified) including fludarabine IV on days -5 to -3 and cyclophosphamide IV on days -5 to -3 or on days -4 and/or -3. The study PI and the protocol team will choose a chemotherapy regimen, for lymphodepletion prior to the PSCA-CAR T cell infusion (with the exception of cohorts 1 and -1 which will not receive lymphodepletion), based on the research participant's disease type and prior therapies. Patients then receive autologous anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T lymphocytes IV over 10-15 minutes at day 0.
  Interventions: Biological: Autologous Anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T-lymphocytes; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Fludarabine Phosphate

INTERVENTIONS:
Biological: Autologous Anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T-lymphocytes — Given IV
  Other Names: Autologous Anti-PSCA(dCH2)BBz-CAR T-cells; Autologous Anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T-cells; PSCA(dCH2)BBzeta-CAR T-cells
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586

SUMMARY:
This phase I trial studies side effects and best dose of PSCA-chimeric antigen receptor (CAR) T cells in treating patients with prostate stem cell antigen positive (PSCA+) castration resistant prostate cancer that has spread to other places in the body (metastatic). PSCA-CAR T cells are immune cells that have been engineered in the laboratory to kill tumor cells. This is done by using a virus to insert a piece of deoxyribonucleic acid (DNA) into the immune cells that allows them to recognize prostate tumor cells. It is not yet known how well PSCA-CAR T cells works in killing tumor cells in patients with metastatic castration resistant prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Define the safety and tolerability of autologous anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T lymphocytes (PSCA-CAR T cells) in patients with PSCA+ metastatic castration resistant prostate cancer (mCRPC).

II. Define the recommended phase 2 dose (RP2D) of PSCA-CAR T cells in patients with PSCA+ mCRPC.

SECONDARY OBJECTIVES:

I. Assess the expansion and persistence of PSCA-CAR T cells.

II. Assess clinical response based on Prostate Cancer Working Group 3 (PCWG3) criteria.

III. Assess survival outcomes (including biochemical progression free survival [PFS], radiographic PFS and overall survival [OS]).

IV. Assess serum cytokine profiles in peripheral blood pre- and post-therapy. V. Describe the PSCA expression level on tumor cells prior to CAR T cell infusion, and the relationship it may have with disease response and observed toxicities.

EXPLORATORY OBJECTIVES:

I. Characterize the phenotypes and frequencies of immune cell subsets in the peripheral blood pre- and post-therapy.

II. Enumerate and characterize tumor-infiltrating lymphocytes (TILs) pre- and post-therapy.

III. Enumerate and analyze gene expression of circulating tumor cells (CTC) pre- and post-therapy.

IV. Analyze circulating cell-free DNA (cfDNA). V. Determine the immunogenicity of PSCA-CAR T cells.

OUTLINE: This is a dose-escalation study.

Patients may receive lymphodepleting regimen at the discretion of the treating physician including fludarabine intravenously (IV) on days -5 to -3 and cyclophosphamide IV on days -5 to -3 or on days -4 and/or -3. Patients then receive autologous anti-PSCA-CAR-4-1BB/TCRzeta-CD19t-expressing T lymphocytes IV over 10-15 minutes at day 0.

After completion of study treatment, patients are followed up at day 1, every 2 days for up to 14 days, weekly for up to 1 month, every month for up to 1 year, and then annually for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have the ability to understand and the willingness to sign a written informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2 or KPS ≥70%.
* Documented castration resistant prostate cancer (mCRPC) (Note: castration will be defined by a testosterone < 50 ng/dL achieved by orchiectomy or luteinizing hormone-releasing hormone [LHRH] agonist/antagonist therapy)

  * Documented PSCA+ tumor expression as evaluated by City of Hope (COH) Pathology Care
  * Progression of disease manifest by one of the following means during treatment with at least one advanced androgen targeted therapy (e.g., abiraterone or enzalutamide)

    * Rising PSA documented on 2 occasions at least 7 days apart, with absolute increase > 2 ng/dL despite testosterone < 50 OR
    * Radiographic evidence of new metastatic foci on computed tomography (CT) or bone scan, or soft tissue progression by Response Evaluation Criteria in Solid Tumors (RECIST)
* Prior chemotherapy with cabazitaxel and/or docetaxel is allowed but not required. If there has been prior chemotherapy, at least 2 weeks must have elapsed prior to leukapheresis
* Prior radiotherapy is allowed provided it was not administered to the only evaluable site of disease and was > 14 days prior to leukapheresis
* No known contraindications to leukapheresis, steroids or tocilizumab
* Total serum bilirubin =< 2.0 mg/dL (to be performed within 42 days of signing the main study consent)

  * Patients with Gilbert syndrome may be included if their total bilirubin is =< 3.0 x upper limit of normal (ULN) and direct bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST) < 5 x ULN (to be performed within 42 days of signing the main study consent)
* Alanine aminotransferase (ALT) < 5 x ULN (to be performed within 42 days of signing the main study consent)
* Creatinine clearance of >= 50 mL/min per the Cockcroft-Gault formula (to be performed within 42 days of signing the main study consent)
* Cardiac function (12 lead-electrocardiography [ECG]) without acute abnormalities requiring investigation or intervention (to be performed within 42 days of signing the main study consent)
* Left ventricular ejection fraction > 40% (to be performed within 42 days of signing the main study consent)
* Participants of reproductive potential must agree to use acceptable birth control methods throughout study therapy and for 3 months after final dose of study treatment

Exclusion Criteria:

* Participants with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of signing the main consent
* Participants with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, including seizure disorder
* History of allergic reactions attributed to compounds of similar chemical or biologic composition or other agents used in this study
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to signing the main consent
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; non-muscle invasive bladder cancer; malignancy treated with curative intent with no known active disease present for >= 3 years
* Uncontrolled active infection
* Active hepatitis B or hepatitis C infection
* Human immunodeficiency virus (HIV) infection
* Any other condition that would, in the investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2026-04-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya B Dorff, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Dorff TB, Blanchard MS, Adkins LN, Luebbert L, Leggett N, Shishido SN, Macias A, Del Real MM, Dhapola G, Egelston C, Murad JP, Rosa R, Paul J, Chaudhry A, Martirosyan H, Gerdts E, Wagner JR, Stiller T, Tilakawardane D, Pal S, Martinez C, Reiter RE, Budde LE, D'Apuzzo M, Kuhn P, Pachter L, Forman SJ, Priceman SJ. PSCA-CAR T cell therapy in metastatic castration-resistant prostate cancer: a phase 1 trial. Nat Med. 2024 Jun;30(6):1636-1644. doi: 10.1038/s41591-024-02979-8. Epub 2024 Jun 12. PMID 38867077

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 (Starting Dose Level 1): 100 million CAR T+ cells
- Dose Level 2 (Dose Level 1b): 100 million CAR T+ cells plus lymphodepletion
  Cyclophosphamide: 500 mg/m2 Given IV
  Fludarabine: 30 mg/m2 Given IV
- Dose Level 3 (Dose Level 1d): 100 million CAR T+ cells plus modified lymphodepletion
  Cyclophosphamide: 300 mg/m2 Given IV
  Fludarabine: 30 mg/m2 Given IV
Period: Overall Study
Arm/Group | Dose Level 1 (Starting Dose Level 1) | Dose Level 2 (Dose Level 1b) | Dose Level 3 (Dose Level 1d)
Started | 3 | 6 | 5
Completed | 3 | 6 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (Starting Dose Level 1) | Dose Level 2 (Dose Level 1b) | Dose Level 3 (Dose Level 1d) | Total
Number analyzed (Participants) | 3 | 6 | 5 | 14
Age, Continuous [Median (Full Range); unit: years] | 62 [59 to 69] | 70 [42 to 73] | 69 [62 to 72] | 69 [42 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 3 | 6 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 3 | 6 | 3 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 5 | 14
Baseline PSA (Prostate Specific Antigen) [Median (Full Range); unit: ng/mL] | 16.5 [10.7 to 20.4] | 88.0 [11.7 to 590.2] | 235.3 [1.8 to 3260.0] | 88.0 [1.8 to 3260.0]

OUTCOME MEASURES:

1. Primary Outcome: Grade 3 Toxicity Profile
Description: Grade 3 toxicity profile as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5 and modified Cytokine Release Syndrome (CRS) grading as applicable post chimeric antigen receptor (CAR) T cell infusion.
Time Frame: Up to 32 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (Starting Dose Level 1) | Dose Level 2 (Dose Level 1b) | Dose Level 3 (Dose Level 1d)
Number analyzed (Participants) | 3 | 6 | 5
Participants
  Anemia : Yes | 2 | 2 | 0
  Anemia : No | 1 | 4 | 5
  Lymphocyte count decreased : Yes | 1 | 0 | 1
  Lymphocyte count decreased : No | 2 | 6 | 4
  Fatigue : Yes | 0 | 2 | 0
  Fatigue : No | 3 | 4 | 5
  Pain : Yes | 0 | 1 | 0
  Pain : No | 3 | 5 | 5
  Cystitis noninfective : Yes | 0 | 2 | 0
  Cystitis noninfective : No | 3 | 4 | 5
  Hematuria : Yes | 0 | 1 | 0
  Hematuria : No | 3 | 5 | 5
  Rash maculo-papular : Yes | 0 | 1 | 0
  Rash maculo-papular : No | 3 | 5 | 5

2. Primary Outcome: Number of Participants Experiencing a Dose-limiting Toxicity (DLT)
Description: Defined by any grade 3 or NCI CTCAE toxicities and modified CRS grading as applicable.
Time Frame: Up to 28 days post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 (Starting Dose Level 1) | Dose Level 2 (Dose Level 1b) | Dose Level 3 (Dose Level 1d)
Number analyzed (Participants) | 3 | 6 | 5
Participants | 0 | 2 | 0

3. Secondary Outcome: Percent of Participants With CAR T Cells Persistence at Day 28
Description: Persistence is defined as CAR T cells comprising at least 7.5 copies/ug of DNA of total CD3 cells.
Time Frame: Days 28 post infusion
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Dose Level 1 (Starting Dose Level 1) | Dose Level 2 (Dose Level 1b) | Dose Level 3 (Dose Level 1d)
Number analyzed (Participants) | 3 | 6 | 5
Percent of participants | 66 [9 to 99] | 66 [22 to 96] | 60 [15 to 95]

4. Secondary Outcome: Expansion of CAR T Cells
Description: Peak expansion (max log10 copies/ug of genomic deoxyribonucleic acid [DNA]) will be described.
Time Frame: Up to 28 days post treatment
Measure: Mean (95% Confidence Interval); unit: log10 copies/ug of DNA
Arm/Group | Dose Level 1 (Starting Dose Level 1) | Dose Level 2 (Dose Level 1b) | Dose Level 3 (Dose Level 1d)
Number analyzed (Participants) | 3 | 6 | 5
log10 copies/ug of DNA | 2.1 [1.6 to 2.6] | 3.3 [2.5 to 4.0] | 2.8 [2.3 to 3.4]

5. Secondary Outcome: Percent of Participants Achieving Stable Disease
Description: Rates and associated 90% Clopper and Pearson binomial confidence limits will be estimated for response based on Prostate Cancer Working Group 3 (PCWG3) criteria.
Time Frame: Up to 1 year post treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level 1 (Starting Dose Level 1) | Dose Level 2 (Dose Level 1b) | Dose Level 3 (Dose Level 1d)
Number analyzed (Participants) | 3 | 6 | 5
percentage of participants | 0 [0 to 71] | 67 [22 to 96] | 60 [15 to 95]

6. Secondary Outcome: Percent of Participants Alive at Six Months
Description: Rates and associated 95% exact Clopper and Pearson binomial confidence intervals will be estimated.
Time Frame: From CAR T cell infusion to death from any cause or last contact date, assessed up to 6 months
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Level 1 (Starting Dose Level 1) | Dose Level 2 (Dose Level 1b) | Dose Level 3 (Dose Level 1d)
Number analyzed (Participants) | 3 | 6 | 5
Percentage of participants | 33 [1 to 91] | 67 [22 to 96] | 40 [5 to 85]

ADVERSE EVENTS:
Time Frame: While on study, up to 3 years
Arm/Group | Dose Level 1 (Starting Dose Level 1) | Dose Level 2 (Dose Level 1b) | Dose Level 3 (Dose Level 1d)
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/6 | 5/5
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/6 | 4/5
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (Starting Dose Level 1) (N=3) | Dose Level 2 (Dose Level 1b) (N=6) | Dose Level 3 (Dose Level 1d) (N=5)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Generalized edema (General disorders) | 1 | 0 | 0
CRS (Immune system disorders) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (Starting Dose Level 1) (N=3) | Dose Level 2 (Dose Level 1b) (N=6) | Dose Level 3 (Dose Level 1d) (N=5)
Anemia (Blood and lymphatic system disorders) | 3 | 6 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 4 | 4
Blurred vision (Eye disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 2 | 2 | 0
Eye pain (Eye disorders) | 0 | 3 | 1
Photophobia (Eye disorders) | 0 | 2 | 0
Periorbital edema (Eye disorders) | 1 | 1 | 1
blepharoconjuctivitis (Eye disorders) | 0 | 1 | 0
corneal abrasion (Eye disorders) | 0 | 1 | 0
left sided subconjuctival hemorrhage (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Ascites (Gastrointestinal disorders) | 1 | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 6 | 3
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1
Fecal incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 5
Vomiting (Gastrointestinal disorders) | 1 | 4 | 1
Chills (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 2 | 6 | 4
Fever (General disorders) | 1 | 3 | 3
Gait disturbance (General disorders) | 0 | 1 | 1
Generalized edema (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 1 | 2
Edema limbs (General disorders) | 1 | 3 | 1
Localized edema (General disorders) | 0 | 3 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 1
CRS (Immune system disorders) | 1 | 2 | 1
Immune reaction (Immune system disorders) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 2 | 0
Papulopustular rash (Infections and infestations) | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 5 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 2 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3 | 0
Alkaline phosphatase increased (Investigations) | 1 | 4 | 3
Aspartate aminotransferase increased (Investigations) | 1 | 4 | 2
Blood bilirubin increased (Investigations) | 0 | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 2 | 1
Cardiac troponin I increased (Investigations) | 0 | 0 | 1
Cardiac troponin T increased (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 1 | 1 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 6 | 5
Lymphocyte count increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 6 | 5
Platelet count decreased (Investigations) | 0 | 3 | 4
Thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0
Weight gain (Investigations) | 2 | 3 | 2
Weight loss (Investigations) | 1 | 4 | 2
White blood cell decreased (Investigations) | 2 | 6 | 5
Ejection fraction decreased (Investigations) | 0 | 1 | 0
Lip sweling (Investigations) | 0 | 0 | 1
night sweats (Investigations) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 4 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 | 2 | 2
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 6 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 4 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 5 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 3 | 2
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 3
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 4 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 1
Irritability (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 2
Hematuria (Renal and urinary disorders) | 2 | 5 | 4
Proteinuria (Renal and urinary disorders) | 2 | 5 | 3
Urinary frequency (Renal and urinary disorders) | 1 | 2 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 2 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 3 | 1
Glucosuria (Renal and urinary disorders) | 0 | 1 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3 | 1
skin tear (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 6 | 5
Hypotension (Vascular disorders) | 0 | 3 | 2
Thromboembolic event (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT03873805/Prot_SAP_000.pdf